CLINICAL TRIAL: NCT00000180
Title: AIT-082 Phase 1B Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0008; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-02

CONDITIONS: Memory Disorders
Keywords: Memory; Mild cognitive impairment; Nerve growth factors
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction | interventions — 4-((3-(1,6-dihyro-6-oxo-9H-purin-9-yl)-1-oxopropyl)amino)benzoic acid

INTERVENTIONS:
Drug: AIT-082

SUMMARY:
AIT-082 is a novel small molecule that crosses the blood-brain barrier to enhance nerve function by increasing levels of neurotrophic growth factors and encouraging nerve sprouting in the brain. Preclinical studies in animals have shown that AIT-082 improves memory in aged animals and in animals with neurological deficits.

This study was a double-blind placebo-controlled safety study that was designed to study whether AIT-082 may delay age-related mental decline. Eight healthy older volunteers at two clinical sites were given single, weekly, rising doses of AIT-082 or placebo for 5 weeks; were tested for side effects and absorption; and underwent a battery of neuropsychological memory tests, including word and number recall tests.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grundman, M.D., M.P.H., Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - Indiana University Alzheimer's Center, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri

REFERENCES:
- [Result] Grundman M, Capparelli E, Kim HT, Morris JC, Farlow M, Rubin EH, Heidebrink J, Hake A, Ho G, Schultz AN, Schafer K, Houston W, Thomas R, Thal LJ; Alzheimer's Disease Cooperative Study. A multicenter, randomized, placebo controlled, multiple-dose, safety and pharmacokinetic study of AIT-082 (Neotrofin) in mild Alzheimer's disease patients. Life Sci. 2003 Jun 20;73(5):539-53. doi: 10.1016/s0024-3205(03)00320-5. PMID 12770610